CLINICAL TRIAL: NCT01233895
Title: Open Label Study of the Anti Insulin-like Growth Factor 1 Receptor (IGF-1R) Monoclonal Antibody, AVE1642, as Single Agent (Dose Escalation, Part 1) and in Combination With Velcade® (Combination, Part 2) in Patients With Recurrent, Refractory Multiple Myeloma (MM)
Brief Title: Study of AVE1642 Anti-IGF1R Monoclonal Antibody in Patients With Advanced Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED6420; AVE1642A/1001 (Other: other sanofi-aventis reference)
Record Dates: First submitted 2010-10-29; First posted 2010-11-03 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — AVE1642; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVE1642/ AVE1642 with Velcade (Experimental)
  Interventions: Drug: AVE1642; Drug: Velcade

INTERVENTIONS:
Drug: AVE1642 — For Part 1, AVE1642 was administered on Day 1 and then every three weeks intra-venously with the dose escalation step starting at 3 mg/kg/infusion with a classical dose escalation schema of 3+3. For Part 2, AVE1642 was administered at doses ranging from 0.5 mg/kg to 12 mg/kg
Drug: Velcade — For Part 2 ONLY, fixed dose of 1.3 mg/m² administered on Days 1, 4, 8, and 11.
  Other Names: Bortezomib

SUMMARY:
Primary Objectives:

Study Part 1: Determine the selected dose of AVE1642 administered every 3 weeks based on pharmacokinetic (PK) (Clearance of AVE1642), pharmacodynamic (PD) (insulin-like growth factor 1 [IGF-1] serum level) parameters, and eventual dose limiting toxicities (DLTs) in patients with recurrent, refractory multiple myeloma (MM).

Study Part 2: Assess the safety of the combination of the selected dose of AVE1642 with the recommended dose of Velcade®.

Secondary Objectives :

Study Part 1:

* To assess the safety profile: type, incidence and intensity of drug related adverse events (AEs)
* To assess the biological activity of AVE1642 (saturation of the receptors and down-regulation) on malignant plasma cells and on peripheral blood mononuclear cells (PBMC) and granulocytes
* To assess the biological activity of AVE1642 on the signalization pathway of the IGF-1 system (phosphorylated akt [pAkt], phosphorylated erk [pErk]) on malignant plasma cells when technically possible
* To define PK profile of AVE1642, and its PD effects on serum IGF 1, GF 2 and IGFBP-3
* To assess clinical efficacy (complete response [CR], partial response [PR], minimal response [MR] and stabilization) based on the European group for Blood and Marrow Transplantation (EBMT) criteria, when possible
* To assess potential immunogenicity by detection of human antihumanized antibodies (HAHA) anti-AVE1642

Study Part 2:

* To detect any PK or PD interaction between AVE1642 and Velcade®
* To assess clinical efficacy (CR, PR, MR, no change [NC]) according to EBMT criteria when appropriate
* To assess biological activity of AVE1642 in combination with Velcade® on malignant plasma cells collected from bone marrow aspirates: saturation and down-regulation of the insulin-like growth factor 1 receptor (IGF-1R) and activity on the signalization pathway of the IGF-1 system (pAkt, pErk) when feasible
* To detect immunogenicity reaction (HAHA)
* To characterize PK and PD profile of a low dose (0.5 mg/kg) of AVE1642 expected to be non biologically active

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma confirmed by bone marrow aspirate or biopsy
* Patient had to have relapsed and/or refractory multiple myeloma after at least 1 standard therapy, and have demonstrated disease progression
* Previous exposure to Velcade was allowed, provided no DLTs of Grade 3 or above had been observed during previous treatment (for Part 2 of the study only)

Exclusion Criteria:

* Prior therapy with any IGF-1 system targeting compound
* History of allogenic stem cell transplantation in case of concomitant immunosuppressive therapy within 6 months before study entry. Patients having undergone autologous stem cell transplantation(s) may have been included in the study
* History of organ transplant and any patient receiving long term systemic immunosuppressive therapy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
definition of the Selected Dose (SD) | 2 years
  Selected Dose will be based on the AVE1642 clearance /IGF-1 plateaus and on safety (less than 33% of pts with dose limiting toxicity (DLT)when administered as single agent in a first part of the study. The safety and pharmacokinetics of the regimen in combination with bortezomib will be assessed in the second part of the study

SECONDARY OUTCOMES:
Assess the efficacy (complete, partial, minimal responses and stabilizations) | 2 years
  According to the European Group for Blood and Marrow Transplantation (EBMT) criteria when appropriate (e.g. baseline M Protein, % Plasma Cells in Bone Marrow,skeletal disease status and at least one evaluable post-baseline assessment)
Pharmacokinetic drug interaction between AVE1642 and Velcade (part 2) | Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- France (3):
  - Sanofi-Aventis Investigational Site Number 250002, Lille
  - Sanofi-Aventis Investigational Site Number 250001, Nantes
  - Sanofi-Aventis Investigational Site Number 250003, Vandœuvre-lès-Nancy
- Sanofi-Aventis Investigational Site Number 380001, Torino, Italy